CLINICAL TRIAL: NCT07045506
Title: Estimating Umbilical Venous Catheter Insertion Depth in Newborns Using Weight or Body Measurements: A Multicenter Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Fawzy Kamel Abdelhamid, Consultant Neonatology, King Fahad Medical City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-542
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Estimating Umbilical Venous Catheter Insertion Depth in Newborns Using Weight or Body Measurements
Keywords: umbilical venous catheter ( UVC) , catheter placement, Gupta method, birth weight-based formula, neonatal intensive care unit, clinical trial,

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 UVC insertion depth estimated using the Umbilicus to Nipple distance (UN) minus 1 (Active Comparator): Neonates who met the eligibility criteria were randomly assigned to one of two groups. Group 1 had their UVC insertion depth estimated using the Umbilicus to Nipple distance (UN) minus 1 cm formula (Gupta method), while Group 2 used the birth weight formula (3*wt +9)/2 (modified Shukla). Randomization was achieved using a computer-generated sequence, with allocation in blocks of four. The neonates were randomized in a 1:1 ratio. Initially, 184 infants were assessed for eligibility to participate in the study. Of these, 4 were excluded due to refusal to participate. The remaining 180 infants were randomly assigned to one of two intervention groups (the Gupta group or the modified Shukla group) in a 1:1 ratio. All infants in both groups received the allocated intervention, with no cases lost to follow-up or discontinuation of the intervention.
  Interventions: Other: UVC insertion
- Group 2 UVC insertion used the birth weight formula (3*wt +9)/2 (modified Shukla) (Active Comparator): Neonates who met the eligibility criteria were randomly assigned to one of two groups. Group 1 had their UVC insertion depth estimated using the Umbilicus to Nipple distance (UN) minus 1 cm formula (Gupta method), while Group 2 used the birth weight formula (3*wt +9)/2 (modified Shukla). Randomization was achieved using a computer-generated sequence, with allocation in blocks of four. The neonates were randomized in a 1:1 ratio. Initially, 184 infants were assessed for eligibility to participate in the study. Of these, 4 were excluded due to refusal to participate. The remaining 180 infants were randomly assigned to one of two intervention groups (the Gupta group or the modified Shukla group) in a 1:1 ratio. All infants in both groups received the allocated intervention, with no cases lost to follow-up or discontinuation of the intervention.
  Interventions: Other: UVC insertion

INTERVENTIONS:
Other: UVC insertion — UVC insertion was performed under sterile conditions according to the unit protocol by a senior NICU physician. For preterm deliveries, written informed consent was obtained from a parent before enrollment in the study. In emergency cases, where the neonate required immediate UVC insertion upon admission to the NICU, a waiver of informed consent was applied. In such instances, parents were informed as soon as possible about their infant's participation in the study, provided with written information, and asked for their consent to include their infant's data in the analysis, with the option to give consent via telephone if they were unable to be present in person.
  After UVC insertion, anteroposterior and lateral thoracoabdominal radiographs were performed to verify the position of the UVC tip.

SUMMARY:
Introduction: The current methods for estimating umbilical venous catheter (UVC) insertion depth, including the umbilical to nipple (Gupta) and the birth weight-based (modified Shukla) formula, have varying accuracy rates.

Objectives: To compare the accuracy of UVC insertion length using the birth weight-based formula versus the surface measurement formula in determining the optimal UVC tip position.

Methods: A multicenter randomized clinical trial was conducted in the neonatal intensive care units (NICUs) of the Second Cluster in Al Riyadh (AL Yamama Hospital and King Fahad Medical City), King Salman Armed Forces Hospital in the Northwestern Region, Tabuk City, Saudi Arabia. Neonates requiring UVC insertion during their NICU admission were randomly assigned to one of two formulas: 1) the umbilicus to nipple distance in centimeters minus 1 (UN - 1) or 2) the modified Shukla weight-based formula in centimeters (3 × birth weight in kg + 9, divided by 2) to estimate the pre-insertion UVC depth and to determine the UVC tip position anteroposterior and lateral thoracoabdominal radiographs were taken and reviewed by a neonatologist, who was blinded to the group assignments. Data analysis was conducted using appropriate statistical methods, ensuring adherence to ethical standards.

DETAILED DESCRIPTION:
I.Project Summary In this randomized clinical study, who are hospitalize in the neonatal intensive care unit pediatric department of King Salman Armed Forces Hospital Northwestern Region KSA Neonates who require umbilical venous catheter (UVC) insertion during their NICU admission will be randomized to one of the 2 formulas 1) umbilicus to the nipple in cm minus 1 (UN - 1) or 2) and birth weight based formula (1.5×birth weight (Kg) + 5.6) for estimation of the pre-insertion UVC depth. UVC will be inserted under sterile condition as per our unit protocol. Then to determine the UVC tip position, anteroposterior and lateral a thoracoabdominal radiograph will be taken.

II.Introduction Umbilical vessel catheterization of newborns was used for more than 60 years (1,2).The ideal position of UVC tip to decrease complications is outside the heart at the junction of inferior vena cava and right atrium (3). UVC related complications are mainly due to catheter malposition as pericardial effusions , cardiac tamponade and cardiac thrombus have been reported with UVCs whose tips lay within the heart (4). There is no definite rule describe how far umbilical catheters should be inserted in the umbilical vein; different methods including the Dunn method, Shukla-Ferrara, modified Shukla-Ferrara and umbilicus to the nipple formulae are used (5). Selection of the most correct methods is very important in terms of decreasing th risk and frequency of complications (6,7). IN KFMC NICU and Alyamah NICU and Pediatric department of King Salman Armed Forces Hospital Northwestern Region KSA , the most commonly used method for estimation of UVC insertion length is the birth weight based formula (3× birth weight (Kg) +9)/2. A recent retrospective study reported that 57% accuracy rate with birth weight based formula(8). In our units no audit done for accuracy rate of UVC dependent on birth weight based formula endpoint

The endpoint measurement of UVC tip determined by anteroposterior x ray (12,13) to check where is the tipe of UVC located that is used in our unit

III.Project Objectives

Research Questions: Does the estimating insertion depth using umbilicus to the nipple in cm minus 1 (UN - 1) formula more accurate than a birth weight-derived formula resulted in more correctly placed umbilical venues catheters.

Primary objective: to compare accuracy rate between UVC insertion length estimated by using 1)umbilicus to the nipple distance in cm minus 1 (UN - 1) formula and 2) Shukla's exact birth weight based formula (3× birth weight (Kg) +9)/2to determine optimum UVC tip position compared against the standard accepted level UVC tip at the level of the diaphragm or the upper border of the 9th and the lower border of the 10th thoracic vertebrae (T9-T10) on the anteroposterior and lateral X-ray Secondary objective: to compare the accuracy rate of UVC tip position between two formulae depend on appropriation of baby to gestational age (AGA, SGA, LGA) AGA: appropriate for gestational age (i.e birth weight between 10th and 90th percentile for gestational age); SGA: Small for gestational age (i.e. birth weight <10th percentile for gestational age); LGA: large for gestational age (i.e. birth weight >90th percentile for gestational age)

IV.Literature Survey/Background Insertion of umbilical venous catheters in newborns admitted to hospital in neonatal intensive care units (NICU) who are preterm or have severe morbidity is a commonly used method for Venus access to maintain fluid support , parenteral nutrition ,administration of blood products, , administration of antibiotic , exchange transfusion and investigations, as well as providing emergency intravenous access (9). Ideally, umbilical venous catheters are placed under guidance of imaging methods. However, umbilical venous catheters are placed without any imaging method in emergency cases in NICUs. This leads to frequent occurrence of malposition of UVC (10,11). The commonly used formulas to estimate the depth of umbilical catheter include a birth weight based formula proposed by Shukla and Ferrara and Dunn's shoulder to umbilical length graph. In our units in the neonatal intensive care unit of KFMC / Al Yamamh Hospital KSA , the most commonly used method for estimation of UVC insertion length is the exact birth weight based formula (3× birth weight (Kg) +9)/2)(14). A recent retrospective study reported a distance from base of umbilicus to nipple distance (UN)-1 cm formula consider best and most accurate insertion depth of UVC with accuracy rate of 84% compared with 57% accuracy rate with birth weight based formula(8). In the literature, few studies have compared the two methods in determining how far umbilical catheters should be inserted in the umbilical vein

ELIGIBILITY:
Inclusion Criteria:

* All neonates who require UVC insertion as part of their intensive care during their NICU admission

Exclusion Criteria:

* Any neonate where the UVC is medically contra-indicated like lower limb ischemia, omphalitis, umbilical bleeding, confirmed intra-vascular thrombosis or DIC.

Neonates with hydrops fetalis, abdominal wall defects, congenital diaphragmatic hernia, major congenital heart disease, and declined to participate or insertion of UVC beyand one week .

Max Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Proportion of correctly inserted UVC at optimum catheter tip position for each method | Within 48 Hours

CONTACTS AND LOCATIONS:
Locations (1):
- Second Cluster ( KFMC and Alyamama Hospital ), Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No